CLINICAL TRIAL: NCT04862494
Title: Paediatric Treatment of Diaphragmatic Eventrations in France: Management Strategies and Long-term Results : an Observational Study.
Brief Title: Diaphragmatic Eventration in Children : Evaluation of Care Strategies and Results in the French Cohort.
Acronym: PedDiaVen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-013
Record Dates: First submitted 2021-04-12; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Diaphragmatic Eventration
Keywords: thoracoscopy; laparoscopy; digestive disorders; restrictive syndrom
MeSH Terms: conditions — Diaphragmatic Eventration; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diaphragmatic eventation with medical surveillance: Patients with a diagnosis of diaphragmatic eventration without respiratory or digestive consequences, thus not requiring surgical repair.
  Interventions: Other: clinical surveillance
- diaphragmatic eventration treated with plication: Patients with a diagnosis of diaphragmatic eventration with respiratory or digestive repercussion, requiring surgical repair.
  Interventions: Procedure: diaphragmatic plication

INTERVENTIONS:
Other: clinical surveillance — regular clinical follow up including chest X-rays, pulmonary investigations, etc...
  Groups: diaphragmatic eventation with medical surveillance
Procedure: diaphragmatic plication — plication of a hemidiaphragm, performed via laparoscopy, thoracoscopy (including robot-assisted surgery), or classical thoracotomy
  Groups: diaphragmatic eventration treated with plication

SUMMARY:
A diaphragmatic eventration is an abnormal and permanent elevation of a portion or an entire intact hemidiaphragm. This rare pathology, found in 0.2 - 1 for every 1000 patients in large radiological series, is either congenital or acquired due to phrenic nerve palsy.

Most diaphragmatic eventrations are asymptomatic and discovered thanks to chest x-rays, where the diaphragmatic dome is elevated and visualized above the 4th intercostal space and sometimes up to the clavicle. Computed tomography or magnetic resonance imaging confirms the eventration by visualizing the diaphragmatic muscle distended and intact, unlike a diaphragmatic rupture or hernia.

Surgical indications are usually due to respiratory disorders or visceral repercussions, such as gastric emptying disorders or acute accidents like gastric volvulus. Surgical treatment is a phrenic plication, which can be performed via a lateral thoracotomy (classical approach), thoracoscopy or laparoscopy.

When surgery is not indicated, follow up consists of regular clinical and radiological monitoring.

There is, however, no consensus when it comes to their medical and surgical management due to the very low number of patients per center and per year, and the fact that very few studies specifically address this subject in the literature.

DETAILED DESCRIPTION:
This is a retrospective multicenter descriptive cohort study based on French national healthcare data. The aim of this study is to describe the current trends in management of diaphragmatic eventrations in France in order to indentify potential risk factors for complications and to improve and homogenize practices.

ELIGIBILITY:
Inclusion Criterion:

* Patients of 16 years of age and under at diagnosis with diaphragmatic eventration, treated since 2010 in a pediatric surgery care unit in France.

Exclusion Criterion:

* Patients with a diaphragmatic hernia
* Patient's parents or legual guardian opposed to being included in the study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: National cohort of all pediatric patients diagnosed with or operated for diaphragmatic eventration since January, 1st, 2010, in a pediatric surgical care unit in France. Patients will be devided into non operated and operated patients for outcome comparisons.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
To assess the level of asymptomatic patients diagnosed with diaphragmatic eventration depending on the type of treatment (surgical or not). | Up to 16 years of age. From the date of diagnosis until the date of last check-up, assessed up to 16 years of age
  Asymptomatic patient rate defined as patients presenting without any digestive, respiratory or orthopaedic symptom.

SECONDARY OUTCOMES:
To assess the occurrence of lung disease in patients with non treated diaphragmatic eventrations | Up to 16 years of age. From the date of diagnosis until the date of last check-up, assessed up to 16 years of age
  Objectified by pulmonary function tests (PFTs), carried out according to the ATS/ERS-GLI (American Thoracic Society and European Respiratory Society-Global Lung Initiative) recommendations.
To assess the rate of digestive symptoms in patients with diaphragmatic eventrations. | Up to 16 years of age. From the date of diagnosis until the date of last check-up, assessed up to 16 years of age
  Clinical assessment of digestive symptoms linked to diaphragmatic eventration and/or to diaphragmatic plication, such à GERD, dumping syndrom, digestive occlusion or pain (scored by visual analogic scale).
To assess the occurrence of orthopaedic impact of non treated diaphragmatic eventrations | Up to 16 years of age. From the date of diagnosis until the date of last check-up, assessed up to 16 years of age
  objectified by the deformation of the spine on chest x-ray measured by the Cobb angle.
To assess the severity rate of postoperative complications | Up to 16 years of age. From the date of diagnosis until the date of last check-up, assessed up to 16 years of age
  Description of postoperative complications encountered after diaphragmatic plication, scored with the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Podevin, MD-PhD, Study Director — University Hospital of Angers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heng L, Alzahrani K, Montalva L, Podevin G, Schmitt F; PedDiaVen collaboration group. Congenital Diaphragmatic Eventration: Should we Maintain Surgical Treatment? A Retrospective Multicentric Cohort Study. J Pediatr Surg. 2025 Jan;60(1):161991. doi: 10.1016/j.jpedsurg.2024.161991. Epub 2024 Oct 10. PMID 39442326